CLINICAL TRIAL: NCT05755607
Title: A Multicenter Prospective Randomized Controlled Study of Robot Pancreaticoduodenectomy Versus Laparoscopic Pancreaticoduodenectomy
Brief Title: A Multicenter Prospective Randomized Controlled Study of RPD Versus LPD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of University of South China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: USC-4310-3
Record Dates: First submitted 2023-02-23; First posted 2023-03-06 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-02

CONDITIONS: Pancreatic Cancer; Common Bile Duct Diseases; Periampullary Carcinoma
Keywords: Robot pancreaticoduodenectomy; laparoscopic pancreaticoduodenectomy; randomized controlled trial; Safety and Efficacy
MeSH Terms: conditions — Pancreatic Neoplasms; Common Bile Duct Diseases

STUDY DESIGN:
Intervention Model Description: The key difference in treatment between the two groups is the surgical approach, with the LPD group undergoing laparoscopic-assisted pancreaticoduodenectomy and the RPD group undergoing robotic-assisted pancreaticoduodenectomy, with all treatments remaining the same except for the surgical approach.
Who Masked: Outcomes Assessor
Masking Description: The way of surgery.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- laparoscopic pancreaticoduodenectomy group (Other): The laparoscopic group will perform the surgical procedure using laparoscopic instruments, with three surgeons involved throughout the procedure.
  Interventions: Procedure: laparoscopic pancreaticoduodenectomy
- Robot Pancreaticoduodenectomy (Other): The robotic team will perform the surgery using the latest generation Da Vinci robotic surgical system, with an additional surgeon assisting in the procedure.
  Interventions: Procedure: Robot Pancreaticoduodenectomy

INTERVENTIONS:
Procedure: laparoscopic pancreaticoduodenectomy — The laparoscopic group will perform the surgical procedure using laparoscopic instruments, with three surgeons involved throughout the procedure.
  Arms: laparoscopic pancreaticoduodenectomy group
Procedure: Robot Pancreaticoduodenectomy — The robotic team will perform the surgery using the latest generation Da Vinci robotic surgical system, with an additional surgeon assisting in the procedure.
  Arms: Robot Pancreaticoduodenectomy

SUMMARY:
laparoscopic pancreaticoduodenectomy(LPD) and Robot Pancreaticoduodenectomy (RPD), as two minimally invasive methods of pancreaticoduodenectomy(PD), have obvious advantages over traditional open pancreaticoduodenectomy(OPD) in terms of reducing surgical trauma and hospitalization time, but there are few studies on their perioperative safety and prognostic effects.However, there are few studies on the perioperative safety and prognostic effects of both procedures. In this trial, the perioperative data and prognosis of both procedures were collected and analyzed through a prospective, multicenter approach to investigate the advantages and disadvantages of both procedures.

DETAILED DESCRIPTION:
In this trial, subjects proposed for PD were randomly divided into two groups, LPD and RPD, according to inclusion and exclusion criteria. Patients in both groups were operated and received perioperative management under the same surgical team and were operated according to the standard PD surgical approach. Subsequently, perioperative clinical data and long-term prognostic data of subjects in both groups will be collected and statistically analyzed to explore a better surgical approach.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old
* Preoperative imaging suggested the presence of space occupying in the head of the pancreas, ampullary abdomen, and distal common bile duct tumor lesions to be treated with Pancreaticoduodenectomy
* No distant transfer
* No significant vascular invasion was received

Exclusion Criteria:

* With tumors of other organs
* Patients unable to tolerate anesthesia and operation due to serious abnormalities in functions of heart, lung and other important organs
* Patients found intraoperative peripheral organ metastasis combined with excision of other organs or found intraoperative radical excision could not be performed and underwent palliative drainage surgery or end the surgery
* Preoperative adjuvant therapy was given

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2028-06-01 (Estimated); Study Completion 2031-07-01 (Estimated)

PRIMARY OUTCOMES:
Rate of long-term Survival | 3 years
  Survival will be documented 3 years after surgery

SECONDARY OUTCOMES:
Unplanned re-admission rate after discharge within 30 days | 3 months
  Serious discomfort requiring re-admission within 30 days after discharge will be recorded, and the safety of the surgical method will be evaluated by this indicator
Incidence of postoperative complications | 2 months
  During hospitalization, common complications of pancreaticoduodenectomy, such as postoperative pancreatic fistula, bile leak, gastrojejunostomy leak, and delayed gastric emptying, will be recorded according to the international diagnostic criteria to evaluate the short-term safety of this surgical approach

CONTACTS AND LOCATIONS:
Overall Officials: Guodong Chen, PhD, Study Chair — The First Affiliated Hospital of University of South China

IPD SHARING:
Plan to Share IPD: No